CLINICAL TRIAL: NCT03195179
Title: The Outcomes of Primary Urethral Realignment Versus Suprapubic Cystostomy After Pelvic Fracture Urethral Injury
Brief Title: Primary Urethral Realignment Versus Suprapubic Cystostomy After Pelvic Fracture Urethral Injury
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Jeremy Myers, Associate Professor, University of Utah
Other Study IDs: 00094160
Record Dates: First submitted 2017-06-16; First posted 2017-06-22 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Pelvic Fracture; Urethra Tear; Urethra Injury Male; Trauma; Surgery
Keywords: pelvic fracture urethral injury; urethra; disruption; trauma
MeSH Terms: conditions — Hip Fractures; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Suprapubic tube placement: Standard of care management for men with complete urethral injuries where a Foley catheter fails to be placed will have a suprapubic tube placed to manage the acute urethral injury. This is a standard of care approach and a retrospective review will be done on the patient record to determine outcomes.
- Urethral realignment: Standard of care management for men with complete urethral injuries where a Foley catheter fails to be placed will undergo urethral realignment with a combined antegrade / retrograde approach within 7 days of injury. This is a standard of care approach and a retrospective review will be done on the patient record to determine outcomes.

SUMMARY:
Pelvic fracture urethral injuries (PFUI) occur in up to 10% of pelvic fractures. It remains controversial whether initial urethral realignment after PFUI decreases rates of urethral obstruction and the need for subsequent urethral procedures.

The retrospective record review should determine the utility of acute urethral realignment after PFUI.

DETAILED DESCRIPTION:
A retrospective chart review to compare outcomes between urethral realignment (group 1) and suprapubic tube (SPT) placement (group 2). The comparison will be between two routinely practiced management approaches of urethral injury after pelvic fracture.

Prior studies demonstrate urethral realignment is associated with a 15% to 50% reduction in urethral obstruction, however, it has also been associated with higher rates of incontinence and erectile dysfunction. Our hypothesis is that early realignment of traumatic urethral injuries after pelvic fracture lowers the incidence of complications like urethral strictures and subsequent need for surgeries.

ELIGIBILITY:
Inclusion Criteria:

Men > 18 years old Blunt force trauma Presence of pelvic fracture Urethral injury Inability to pass a Foley catheter retrograde through the injury into the bladder

Exclusion Criteria:

Straddle type urethral injuries without a pelvic fracture Passage of a catheter successfully in a retrograde fashion

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — Pelvic fracture urethral injuries are only treated by this method in men. Female urethral injuries are very rare and most often treated with immediate surgical repair.
Study Population: Men experiencing a traumatic pelvic fracture urethral injury where there is a major urethral disruption that prevents passage of a catheter or a retrograde cystoscope.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Urethral obstruction | Through study completion, an average of 1 year
  Rates of urethral obstruction identified by urethrogram or cystoscopy

SECONDARY OUTCOMES:
Treatment rate for urethral obstruction | Through study completion, an average of 1 year
  The rate of interventions for urethral obstruction after injury
Urethroplasty complexity - gap length during urethroplasty | Through study completion, an average of 1 year
  The gap between the 2 severed ends of the urethra
Urethroplasty complexity - bulbar mobilization length during urethroplasty | Through study completion, an average of 1 year
  The length of bulbar mobilization
Urethroplasty complexity - corporal splitting during urethroplasty | Through study completion, an average of 1 year
  The need to split the 2 corporal bodies
Urethroplasty complexity - total obstruction of the urethra during urethroplasty | Through study completion, an average of 1 year
  Finding the urethra was completely obstructed
Urethroplasty complexity - urethral diverticulum discovered during urethroplasty | Through study completion, an average of 1 year
  Finding a urethral diverticulum
Urethroplasty complexity - urethral fistula present | Through study completion, an average of 1 year
  Finding a urethral fistula
Urethroplasty complexity - inferior pubectomy during urethroplasty | Through study completion, an average of 1 year
  The need to remove the inferior portion of the symphysis pubis
Urethroplasty complexity - total pubectomy during urethroplasty | Through study completion, an average of 1 year
  The need to remove the complete symphysis pubis
Erectile function- SHIM score | Through study completion, an average of 1 year
  Erectile function measured by the Sexual Health Inventory for Men (SHIM)
Erectile function - medical treatment rates | Through study completion, an average of 1 year
  Measured by the need for pharmacologic treatment of erectile dysfunction
Erectile function - surgical treatment rates | Through study completion, an average of 1 year
  Rates of surgical treatment of erectile dysfunction
Incontinence | Through study completion, an average of 1 year
  Rates of surgical treatment of incontinence
Post-injury complications | 3 month period post acute urethral injury
  Calvien-Dindo grading

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Myers, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No